CLINICAL TRIAL: NCT04205448
Title: Early Identification and Intervention in Risk of Falling Among Seniors i Bomlo Municipality
Brief Title: Fall Prevention Study Among Seniors in Bomlo
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kjersti Helen Folleso (Other)
Responsible Party: Sponsor-Investigator, Kjersti Helen Folleso, Community physician, Bomlo Municipality
Organization: Bomlo Municipality (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: BK-KS01
Record Dates: First submitted 2019-12-18; First posted 2019-12-19 (Actual); Last update posted 2021-01-28 (Actual); Status verified 2021-01

CONDITIONS: Fall

STUDY DESIGN:
Intervention Model Description: RCT
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercize group (Experimental): 10 weeks of physical exercise. Testing of strength and balance.
  Interventions: Behavioral: Physical exercize
- Control group (No Intervention): Testing of strength and balance.

INTERVENTIONS:
Behavioral: Physical exercize — 10 weeks group exercize followed by community-based voluntary exercize
  Arms: Exercize group

SUMMARY:
Recruiting seniors age 65-85 at risk of falling in Bomlo municipality. Clinical tests performed by physiotherapist. If risk of falling is confirmed, participants will be randomized to either intervention group with fall-preventing exercize program or to a control group. Follow-up over 5 years.

DETAILED DESCRIPTION:
Participants randomized to either exercise group or control group. Tests for balance and strength performed by physiotherapist at inclusion, and after three and six months and one year for both groups. Further follow-up and further inclusion of participants had to be terminated due to the pandemic in Mach 2020, when group activities were no longer allowed.

ELIGIBILITY:
Inclusion Criteria:

* Age 65-85, home-dwellers in Bomlo municipality, capable of following up group-exercize, informed consent.

Exclusion Criteria:

* Serious illness, in need of walking-aid indoors, moderate to severe cognitive impairment

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2021-01-25 (Actual)

PRIMARY OUTCOMES:
Fall-related injuries | First year
  identified in electronic patient record in primary care

CONTACTS AND LOCATIONS:
Overall Officials: Kjetil A Gjoesaeter, Study Chair — Bomlo Municipality
Locations (1):
- Bomlo municipality, Bremnes, Bomlo, Norway

IPD SHARING:
Plan to Share IPD: Yes
Accepted for publication in Norwegian scientific journal "Utposten".
Supporting Information: Study Protocol, CSR
Time Frame: Spring 2021
Access Criteria: Open access, available in Norwegian
URL: http://www.utposten.no